CLINICAL TRIAL: NCT04908514
Title: A Multi-Center, Open-Label, Phase 2 Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of ADX-629 Administered Orally to Subjects With Plaque Psoriasis
Brief Title: A Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADX-629-PS-001
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-01

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — ADX-629

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADX-629 250 mg administered orally twice daily (BID) for approximately 12 weeks. (Experimental)
  Interventions: Drug: ADX-629

INTERVENTIONS:
Drug: ADX-629 — ADX-629 administered orally twice daily (BID) for approximately 12 weeks.

SUMMARY:
A Multi-Center, Open-Label, Phase 2 Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of ADX-629 Administered Orally to Subjects with Plaque Psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female 18 years of age or older.
* Subject has provided written informed consent.
* Females must be post-menopausal, surgically sterile, or use a highly effective method of birth control during the trial and for 30 days after the last administration of test article. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at Visit 1/Screening and Visit 2/Baseline.
* Male subjects who are not surgically sterile (e.g., vasectomy performed at least 6 months prior to trial entry) and are sexually active with a female partner who is of childbearing potential must agree to use an effective form of birth control for the duration of the trial and for 90 days after completion of treatment.
* Subject, in the investigator's opinion, is in good general health and free of any disease state or physical condition that might impair evaluation of plaque psoriasis or exposes the subject to an unacceptable risk by trial participation.

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the trial.
* Subject has a physical condition which, in the investigator's opinion, might impair evaluation of plaque psoriasis or which exposes the subject to an unacceptable risk by trial participation.
* Subject is currently enrolled in an investigational drug, biologic, or device trial.
* Subject has used an investigational drug, investigational biologic, or investigational device treatment within 30 days prior to Visit 2/Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TCR Medical Corporation, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ten subjects were enrolled in the trial.
Groups:
- ADX-629: ADX-629 250mg was administered orally twice daily (BID) for 12 weeks.
Period: Overall Study
Arm/Group | ADX-629
Started | 10
Completed | 7
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- ADX-629: ADX-629 250mg was administered orally BID for 12 weeks.
Arm/Group | ADX-629
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Total Body Surface Area Affected [Mean (Standard Deviation); unit: Percentage (%)] | 19.9 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Psoriasis Area and Severity Index (PASI)
Description: The change from baseline for PASI score was assessed on a 0 to 72 scale (0 = none, 72 = maximum severity). Mixed model for repeated measures (MMRM) analysis was performed using change from baseline as the dependent variable, baseline as a covariate, and visit as a factor.
Time Frame: The efficacy assessment period was baseline, Week 4, Week 8, and Week 12. Baseline was the day prior to randomization.
Population: Safety population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADX-629
Number analyzed (Participants) | 8
score on a scale
  Week 4 | -4.3 (5.2)
  Week 8 | -7.6 (6.9)
  Week 12 | -8.0 (7.5)

2. Secondary Outcome: Number of Subjects With a ≥ 50% Reduction Change From Baseline for PASI Score
Description: The number of subjects with a ≥ 50% reduction change from baseline for PASI score at Week 12 (end of treatment) was assessed on a 0 to 72 scale (0 = none, 72 = maximum severity). MMRM analysis was performed using change from baseline as the dependent variable, baseline as a covariate, and visit as a factor.
Time Frame: The efficacy assessment period was Week 1 - Week 12. Baseline was the day prior to randomization.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-629
Number analyzed (Participants) | 7
Participants | 3

3. Secondary Outcome: Number of Subjects With a ≥ 75% Reduction Change From Baseline for PASI Score
Description: The number of subjects with a ≥ 75% reduction change from baseline for PASI score at Week 12 (end of treatment) was assessed on a 0 to 72 scale (0 = none, 72 = maximum severity). MMRM analysis was performed using change from baseline as the dependent variable, baseline as a covariate, and visit as a factor.
Time Frame: The efficacy assessment period was Week 1 - Week 12. Baseline was Day 1 prior to randomization.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-629
Number analyzed (Participants) | 7
Participants | 2

4. Secondary Outcome: Change From Baseline in the Investigator's Global Assessment (IGA)
Description: The change from baseline for IGA score is based on a five-point scale ranging from 0 to 4 (0 = clear, 4 = severe). MMRM analysis was performed using change from baseline as the dependent variable, baseline as a covariate, and visit as a factor.
Time Frame: The efficacy assessment period was baseline, Week 4, Week 8, and Week 12. Baseline was the day prior to randomization.
Population: Safety population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADX-629
Number analyzed (Participants) | 7
score on a scale
  Week 4 | -0.50 (0.02)
  Week 8 | -0.68 (0.02)
  Week 12 | -0.85 (0.35)

ADVERSE EVENTS:
Time Frame: Approximately 12 weeks
Arm/Group | ADX-629
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADX-629 (N=10)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT04908514/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT04908514/SAP_001.pdf